CLINICAL TRIAL: NCT05726019
Title: Colchicine in Patients Undergoing Coronary Artery Bypass Grafting After Acute Coronary Syndrome: an Open-label Randomized Trial
Brief Title: Colchicine in Patients Undergoing Coronary Artery Bypass Grafting After Acute Coronary Syndrome
Acronym: COCAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SDC 5302/21/077
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; Coronary Artery Bypass; Myocardial Reperfusion; Postpericardiotomy Syndrome; Postoperative Atrial Fibrilation; Perioperative Myocardial Infarction
Keywords: Colchicine; Acute Coronary Syndrome; Coronary Artery Bypass; Myocardial Reperfusion; Postpericardiotomy Syndrome; Postoperative atrial fibrilation; Perioperative Myocardial Infarction; Coronary Artery Disease; Atherosclerosis; Cardiac Surgery; Cardiology
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Postpericardiotomy Syndrome; Atherosclerosis | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, open-label, randomized study. Patients with acute coronary syndrome, who meet criteria for surgical myocardial revascularization, will be selected and randomize, with drug addition, in the intervention group, within a maximum of 24 hours after randomization and maintained for up to 30 days after coronary artery bypass grafting.
  Inclusion criteria: Individuals with acute coronary syndrome, with indication for myocardial revascularization surgery, of both genders, aged over 18 years.
  Exclusion criteria: Inability to sign the informed consent form; Current use of colchicine; Current use of long-term corticosteroid therapy; Inflammatory bowel disease or chronic diarrhea; Clinically significant non-transient haematological abnormalities; Renal dysfunction, with creatinine greater than 2 times the upper limit of normality; Severe liver disease; Drug addiction or alcoholism; History of clinically significant sensitivity to colchicine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Active Comparator): Oral tablet colchicine 0.5mg, twice a day, will be started within 24 hours after randomization and maintained until 30 days after coronary artery bypass grafting.
  Interventions: Drug: Colchicine
- Conventional treatment (No Intervention): The control group will follow conventional treatment guided by current guidelines.

INTERVENTIONS:
Drug: Colchicine — Oral tablet colchicine 0.5mg, twice a day, will be started within 24 hours after randomization and maintained until 30 days after coronary artery bypass grafting.
  Arms: Colchicine

SUMMARY:
The present study seeks to evaluate the effectiveness of the use of perioperative colchicine with regard to operative complications, in patients with acute coronary syndrome and indication for cardiac post-surgical revascularization.

Patients will be selected and randomized while still in the emergency room and medication (colchicine 0.5mg every 12 hours or placebo) will be started within 24 hours of randomization, being maintained for 30 days after surgery.

DETAILED DESCRIPTION:
Atherosclerotic disease and its consequences, such as cardiovascular and cerebrovascular disease, are the main causes of morbidity and mortality worldwide, with a rising prevalence as the age pyramid changes with the advancement of society's modernization and medical development. Despite advances, the risk of a new cardiovascular event persists in patients with acute coronary syndrome at around 20% in 3 years.

The search for intervention in the inflammatory pathway of atherosclerotic disease in acute coronary syndrome has been the subject of several studies in recent years. In particular, colchicine, a low-cost medication that acts on the inflammatory, atherosclerotic and arrhythmic process, has been the subject of studies in the setting of acute and chronic coronary syndrome and in the perioperative period of coronary artery bypass grafting.

In the elective perioperative context, it presents data that point to a reduction in myocardial injury and post-pericardiotomy syndrome. In addition to the pathophysiological therapeutic potential in postoperative atrial fibrillation, despite not having been demonstrated in a clinical study.

The present study seeks to evaluate the effectiveness of the use of perioperative colchicine with regard to operative complications, in patients with acute coronary syndrome and indication for cardiac post-surgical revascularization.

Patients will be selected and randomized while still in the emergency room and medication (colchicine 0.5mg every 12 hours or placebo) will be started within 24 hours of randomization, being maintained for 30 days after surgery.

The primary outcome will be a composite of postpericardiotomy syndrome, postoperative fibrillation, and periprocedural infarction. Secondary outcomes will be: (1) Death; (2) acute myocardial infarction; (3) stroke; (4) Readmission; (5) Post-pericardiotomy syndrome; (6) Postoperative atrial fibrillation; (7) Periprocedural infarction; (8) Infection; (9) myocardial injury; (10) Length of stay.

Evidences on the use of colchicine in the perioperative scenario of myocardial revascularization in patients with acute coronary syndrome are scarce, and the present study is a pioneer in this evaluation.

Objective documentation of the benefit of colchicine would imply the prescription of the current medication, with great potential for modifying the guidelines of specific medical societies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute coronary syndrome, with indication for myocardial revascularization surgery
* Patients of both genders, aged over 18 years.

Exclusion Criteria:

* Inability to sign the informed consent form;
* Current use of colchicine;
* Current use of long-term corticosteroid therapy
* Inflammatory bowel disease or chronic diarrhea;
* Clinically significant non-transient haematological abnormalities;
* Renal dysfunction, with creatinine greater than 2 times the upper limit of normality;
* Severe liver disease;
* Drug addiction or alcoholism;
* History of clinically significant sensitivity to colchicine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-05 (Actual); Primary Completion 2025-02-05 (Estimated); Study Completion 2025-02-05 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of postpericardiotomy syndrome, postoperative fibrillation, and periprocedural myocardial infarction. | 30 days after coronary artery bypass graft

SECONDARY OUTCOMES:
Death | 30 days after coronary artery bypass graft
Myocardial infarction | 30 days after coronary artery bypass graft
Stroke | 30 days after coronary artery bypass graft
Hospital readmission | 30 days after coronary artery bypass graft
Postpericardiotomy syndrome | 30 days after coronary artery bypass graft
Postoperative fibrillation | 30 days after coronary artery bypass graft
Periprocedural myocardial infarction | 30 days after coronary artery bypass graft
Infection | 30 days after coronary artery bypass graft
  Infection of any kind
Myocardial injury | 30 days after coronary artery bypass graft
Length of stay | 30 days after coronary artery bypass graft

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute - University of São Paulo, São Paulo, São Paulo, Brazil